CLINICAL TRIAL: NCT07399080
Title: Real-World Clinical Outcomes of GENOSS PCB (Paclitaxel-coated Balloon) for Femoropopliteal Artery Disease: A Prospective, Multicenter, Observational Study
Brief Title: Clinical Outcomes of GENOSS PCB for Femoropopliteal Artery Disease
Acronym: GENOSS PCB
Status: Enrolling by invitation | Type: Observational
Sponsor: Genoss Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-DS1411-1
Record Dates: First submitted 2025-09-30; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-08

CONDITIONS: PTA (Percutaneous Transluminal Angioplasty ); Femoropopliteal Artery Disease
MeSH Terms: conditions — Truncus Arteriosus, Persistent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GENOSS® Peripheral DCB PTA Catheter: Patient treated with GENOSS PCB in the femoropopliteal artery disease

SUMMARY:
The GENOSS PCB study aims to evaluate the safety and efficacy of a Paclitaxel-coated PTA Balloon Catheter(GENOSS® PCB) in patients with the femoropopliteal artery disease.

DETAILED DESCRIPTION:
This prospective, open-label, multicenter, observational study will enroll patients with femoropopliteal artery disease undergoing PTA with the GENOSS® PCB at 10 hospitals.

Because this is an observational study, the number of participants will not be calculated separately, but a total of 200 participants are planned to be recruited during the study period.

All patients will be followed up at 12 months postprocedure to evaluate the safety and efficacy of the paclitaxel-coated PTA balloon catheter.

ELIGIBILITY:
<Inclusion criteria>

Enrollment in the study was limited to patients who met the following inclusion criteria:

1. Subject was ≥19 years of age.
2. Subject had target limb Rutherford classification 2, 3, 4 or 5.
3. Subject with femoropopliteal artery disease who underwent percutaneous transluminal angioplasty using the GENOSS PCB.
4. At least one patent native ouflow artery to the ankle of foot, free from significant stenosis (≥50% stenosis) as confirmed by angiography.
5. Subject provided written informed consent and was willing to comply with the study follow-up requirements.

<Exclusion criteria>

Patients were not permitted to enroll in the study if they met any of the following exclusion criteria:

1. Subjects was allergic to paclitaxel.
2. Subjects with contraindications or hypersensitivity to antiplatelet therapy.
3. Subject had life expectancy of less than 2 years.
4. Women who were pregnant, breast-feeding or intended to become pregnant.
5. Subject was participating in another investigational drug or medical device study.
6. Subject was unwilling or unable to comply with procedures specified in the protocol or had difficulty or inability to return for follow-up visits as specified by the protocol.

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with percutaneous transluminal angioplasty with GENOSS® PCB in the femoropopliteal artery disease
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
The primary safety endpoint | at 12 months post procedure
  The primary safety endpoint is the Major Adverse Events (MAEs)-free rate, defined as a composite of freedom from all-cause death through 1month post procedure and/or freedom from both major target limb amputation and/or clinically-driven target lesion revascularization (TLR) through 12months post procedure.
The primary effectiveness endpoint | at 12 months post procedure
  The primary effectiveness endpoint is a primary patency, defined as a composite of freedom from clinically driven target lesion revascularization (CD-TLR) and freedom from binary restenosis (restenosis defined as peak systolic velocity ratio [PSVR] ≥ 2.4 assessed by duplex ultrasound or ≥ 50% stenosis as assessed by CT angiography) through 12months post procedure.

SECONDARY OUTCOMES:
Target lesion revascularization (TLR, %) | at 1 month, 6 months, and 12 months post procedure
  defined as any re-intervention within the target lesion due to symptoms or drop of ABI/TBI of ≥ 20% or > 0.15 when compared to post procedure baseline.
Change in Rutherford classification | at 1 month, 6 months, and 12 months post procedure
  Clinical improvement as assessed by changes in target limb Rutherford classification from baseline.
Change in ABI (Ankle-brachial index) (or TBI (Toe-brachial index)) | at 1 month, 6 months, and 12 months post procedure
  Change in ABI (ankle-brachial index) from baseline
Device success rate | during the procedure
  defined as successful delivery, balloon inflation and deflation and retrieval of the intact study device without burst below the rated burst pressure (RBP).
Procedural success rate (%) | immediately post procedure
  defined as residual stenosis of ≤ 50% by core laboratory.
Clinical success | up to 1 week
  Clinical success is defined as procedural success without complications (i.e. death, major target limb amputation, clinically-driven TLR) during the hospital stay post procedure.
All-cause death (%) | at 12 months post procedure
Target vessel revascularization (TVR, %) | at 1 month, 6 months, and 12 months post procedure
Major target limb amputation (%) | at 12 months post procedure
  defined as any amputation above the ankle on the target limb.

CONTACTS AND LOCATIONS:
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided